CLINICAL TRIAL: NCT04952818
Title: Radiomics Based on Preoperative Imaging of Giant Cell Tumor of the Spine to Predict the Early Recurrence and Survival of Giant Cell Tumor of the Spine After Surgery, and the Expression Levels of P53, VEGF, RANK, RANKL and Other Prognostic-related Molecular Markers.
Brief Title: The Value of Preoperative Diagnosis and Prognostic Prediction Based on Radiomics of Giant Cell Tumor of Spine
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019460
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2019-08

CONDITIONS: Spinal Tumor
Keywords: giant cell tumor of bone; radiomics; recurrence; spine tumor
MeSH Terms: conditions — Spinal Cord Neoplasms; Giant Cell Tumor of Bone; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RANK/RANKL low expression
  Interventions: Diagnostic Test: RANK/RANKL(RANK: Receptor Activator of Nuclear factor Kappa-Β /RANKL:Receptor Activator of Nuclear factor Kappa-Β Ligand)
- RANK/RANKL high expression
  Interventions: Diagnostic Test: RANK/RANKL(RANK: Receptor Activator of Nuclear factor Kappa-Β /RANKL:Receptor Activator of Nuclear factor Kappa-Β Ligand)

INTERVENTIONS:
Diagnostic Test: RANK/RANKL(RANK: Receptor Activator of Nuclear factor Kappa-Β /RANKL:Receptor Activator of Nuclear factor Kappa-Β Ligand) — Immunohistochemical staining was performed using the following antibodies: anti-RANK antibody from Bioss Company (No.bs-2695R) and anti-RANKL antibody from Abcam (No.ab222215).

SUMMARY:
1. Exploit CT (plain scan), enhanced CT and fMRI based radiomic biomarkers, explore their correlation with the prognostic molecular markers of spinal GCTB(p53/vegf/rank/rankl…), and help accurate diagnosis of GCTB.
2. Exploring a new method of preoperative risk stratification for spinal GCTB, and establishing radiomic model combined with clinical features. Exploring the GCTB biological behavior prediction model and the prognosis prediction of GCTB.

DETAILED DESCRIPTION:
This study intends to conduct a systematic review of patients with spinal GCTB who have undergone standardized imaging (CT or MRI) in our hospital since 2006 to obtain case samples, conduct standardized clinical and imaging data extraction and analysis, and fully integrate histopathology and clinical follow-up results. To preliminarily explore the value of postoperative imaging-based radiomics markers in the preoperative precise diagnosis of spinal GCTB, risk stratification and prediction of tumor biological behavior.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with spinal GCTB who underwent surgical resection or biopsy without preoperative chemotherapy or radiotherapy were included in this study.

Exclusion Criteria:

* i) The CT scan was performed more than 1 week before surgery ii) Poor image quality. Such as surrounding structure artifacts; iii) The remaining tumor tissue in the postoperative paraffin specimen is too little to be used for reanalysis; iv) Cases with negative H3F3A (H3 histone, family 3A) staining were excluded; v) Incomplete clinical information.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with spinal GCTB
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
RANK/RANKL | 2020
  Grade:low;high(Receptor Activator of Nuclear factor Kappa-Β/Ligand)
VEGF | 2020
  Grade:low;high(Vascular Endothelial Growth Factors)
p53 | 2020
  Grade:low;high(Tumor Suppressor Protein)

SECONDARY OUTCOMES:
Recurrence | 2020
  recurrence group/non-recurrence group

CONTACTS AND LOCATIONS:
Overall Officials: Ning Lang, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University third hospital, Beijing, Please Select An Option Below, China

IPD SHARING:
Plan to Share IPD: No